CLINICAL TRIAL: NCT01441999
Title: Proximal Junctional Kyphosis Following Long Instrumented Spinal Fusion: The Effect of Implant Selection
Acronym: PJK
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: principal investigator decision
Sponsor: Globus Medical Inc (Industry)
Collaborators: University of Michigan (Other); Polaris Spine and Neurosurgery Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RGC11-001
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Kyphosis
Keywords: Rigid rods; less rigid rods; prevent kyphosis; long constructs
MeSH Terms: conditions — Kyphosis

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Less rigid rods (Active Comparator): Titanium rods that have a soft, plastic end
  Interventions: Device: Less rigid rod
- Rigid Rods (Active Comparator): Titanium rods
  Interventions: Device: Rigid Rod

INTERVENTIONS:
Device: Less rigid rod — Titanium rod with semi rigid end
  Other Names: TRANSITION
  Arms: Less rigid rods
Device: Rigid Rod — Rigid Titanium rods
  Other Names: REVERE
  Arms: Rigid Rods

SUMMARY:
The treatment of adult deformity has improved with the development and use of modern segmental instrumentation, including posterior instrumentation. However, the incidence of proximal junctional kyphosis (PJK) caused by the accelerated degeneration of the joint capsules and smaller articular processes in the proximal junctional region has also been noted.

One potential way of decreasing PJK is to decrease the structural rigidity of the construct at the top thereby providing a transition to the non-instrumented spine and allowing for less facet capsule and muscle disruption.

DETAILED DESCRIPTION:
While a possible solution to PJK is to reduce structural rigidity at the top of the construct, there is a need to investigate it. In the proposed study, the investigators will compare the rate of proximal junctional kyphosis in patients treated with a stainless steel rod (REVERE Stabilization System) versus those treated with TRANSITION Stabilization System.

Patient outcome measures (Scoliosis Research Society (SRS-22), SF12 and ODI) and radiographic measurements (including lumbar lordosis (L1-S1), adjacent segment kyphosis, thoracolumbar kyphosis (T10-L2), sagittal balance, sacral slope, and pelvic incidence) will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with degenerative spondylolisthesis with objective evidence of neurologic impairment, kyphosis, and failed previous fusion (pseudoarthrosis) requiring treatment with an instrumented posterior fusion from the thoracolumbar junction (T10-L1) to the sacrum
* At least 18 years of age and maximum 70 years of age
* Ability to provide Informed Consent for study participation and patients to return for all follow-up visits

Exclusion Criteria:

* Presence of systemic or localized infection
* Previous fusion attempt at the involved level(s)
* More than three previous open, posterior, lumbar spinal surgical procedures at the involved level(s)
* Trauma at the levels to be fused
* Previous documentation of osteopenia or osteomalacia
* Diagnosis of a condition or requires postoperative medication(s), which may interfere with bony/soft tissue healing
* Presence of a disease entity or condition which totally precludes possibility of bony fusion (e.g. metastatic cancer, HIV, long term use of steroids, etc.)
* Immunosuppressive disorder
* Pregnancy
* History of alcohol and/or drug abuse
* Any known allergy to a metal alloy
* Mentally incompetent or prisoner
* Currently a participant in another study
* Preoperative structural deformity in the thoracic spine (kyphosis >60 degrees, Coronal curve >40 degrees)
* Circumferential fusion above L1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Evidence of Proximal Junction Kyphosis as determined by radiographic measurements during follow up visits | 2 years
  Radiographs will be taken to measure lumbar lordosis, adjacent segment kyphosis, thoracolumbar kyphosis, sagittal balance, Sacral slope and pelvic incidence.

SECONDARY OUTCOMES:
Patient outcome measures | 2 years
  Forms to be completed at follow up visits will include VAS, SRS 22, SF12, ODI, Patient Satisfaction, Work Status Assessment and Odom's criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Cunningham, PhD, Study Director — Globus Medical Inc
Locations (3):
- United States (2):
  - Peachtree Neurosurgery, Atlanta, Georgia
  - Department of Neurosurgery, University of Michigan, Ann Arbor, Michigan
- Department of Orthopedic Surgery, University of Copenhagen, Denmark, Copenhagen, Denmark

REFERENCES:
- [Background] Glattes RC, Bridwell KH, Lenke LG, Kim YJ, Rinella A, Edwards C 2nd. Proximal junctional kyphosis in adult spinal deformity following long instrumented posterior spinal fusion: incidence, outcomes, and risk factor analysis. Spine (Phila Pa 1976). 2005 Jul 15;30(14):1643-9. doi: 10.1097/01.brs.0000169451.76359.49. PMID 16025035
- [Background] Hee HT, Yu ZR, Wong HK. Comparison of segmental pedicle screw instrumentation versus anterior instrumentation in adolescent idiopathic thoracolumbar and lumbar scoliosis. Spine (Phila Pa 1976). 2007 Jun 15;32(14):1533-42. doi: 10.1097/BRS.0b013e318067dc3d. PMID 17572624
- [Background] Hollenbeck SM, Glattes RC, Asher MA, Lai SM, Burton DC. The prevalence of increased proximal junctional flexion following posterior instrumentation and arthrodesis for adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2008 Jul 1;33(15):1675-81. doi: 10.1097/BRS.0b013e31817b5bea. PMID 18580741
- [Background] Kim YJ, Bridwell KH, Lenke LG, Kim J, Cho SK. Proximal junctional kyphosis in adolescent idiopathic scoliosis following segmental posterior spinal instrumentation and fusion: minimum 5-year follow-up. Spine (Phila Pa 1976). 2005 Sep 15;30(18):2045-50. doi: 10.1097/01.brs.0000179084.45839.ad. PMID 16166893
- [Background] Kim YJ, Lenke LG, Bridwell KH, Kim J, Cho SK, Cheh G, Yoon J. Proximal junctional kyphosis in adolescent idiopathic scoliosis after 3 different types of posterior segmental spinal instrumentation and fusions: incidence and risk factor analysis of 410 cases. Spine (Phila Pa 1976). 2007 Nov 15;32(24):2731-8. doi: 10.1097/BRS.0b013e31815a7ead. PMID 18007253
- [Background] Lee GA, Betz RR, Clements DH 3rd, Huss GK. Proximal kyphosis after posterior spinal fusion in patients with idiopathic scoliosis. Spine (Phila Pa 1976). 1999 Apr 15;24(8):795-9. doi: 10.1097/00007632-199904150-00011. PMID 10222531
- [Background] Yang SH, Chen PQ. Proximal kyphosis after short posterior fusion for thoracolumbar scoliosis. Clin Orthop Relat Res. 2003 Jun;(411):152-8. doi: 10.1097/01.blo.0000069885.72909.bb. PMID 12782870
- [Background] Kim YJ, Bridwell KH, Lenke LG, Glattes CR, Rhim S, Cheh G. Proximal junctional kyphosis in adult spinal deformity after segmental posterior spinal instrumentation and fusion: minimum five-year follow-up. Spine (Phila Pa 1976). 2008 Sep 15;33(20):2179-84. doi: 10.1097/BRS.0b013e31817c0428. PMID 18794759
- [Background] Helgeson MD, Shah SA, Newton PO, Clements DH 3rd, Betz RR, Marks MC, Bastrom T; Harms Study Group. Evaluation of proximal junctional kyphosis in adolescent idiopathic scoliosis following pedicle screw, hook, or hybrid instrumentation. Spine (Phila Pa 1976). 2010 Jan 15;35(2):177-81. doi: 10.1097/BRS.0b013e3181c77f8c. PMID 20081513
- [Background] Wang J, Zhao Y, Shen B, Wang C, Li M. Risk factor analysis of proximal junctional kyphosis after posterior fusion in patients with idiopathic scoliosis. Injury. 2010 Apr;41(4):415-20. doi: 10.1016/j.injury.2010.01.001. Epub 2010 Jan 27. PMID 20106476
- [Background] Bunge EM, Juttmann RE, de Kleuver M, van Biezen FC, de Koning HJ; NESCIO group. Health-related quality of life in patients with adolescent idiopathic scoliosis after treatment: short-term effects after brace or surgical treatment. Eur Spine J. 2007 Jan;16(1):83-9. doi: 10.1007/s00586-006-0097-9. Epub 2006 Apr 12. PMID 16609857
- [Background] Taylor TC, Wenger DR, Stephen J, Gillespie R, Bobechko WP. Surgical management of thoracic kyphosis in adolescents. J Bone Joint Surg Am. 1979 Jun;61(4):496-503. PMID 438235
- [Background] Glassman SD, Schwab F, Bridwell KH, Shaffrey C, Horton W, Hu S. Do 1-year outcomes predict 2-year outcomes for adult deformity surgery? Spine J. 2009 Apr;9(4):317-22. doi: 10.1016/j.spinee.2008.06.450. Epub 2008 Sep 6. PMID 18774752